CLINICAL TRIAL: NCT05972577
Title: Optimization of Older Adult Allogeneic Hematopoietic Cell Transplant Candidates to Improve Survival (OTIS)
Brief Title: Geriatric Optimization Plan to Improve Survival in Older Adult Allogeneic Hematopoietic Cell Transplant Candidates, OTIS Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Sarah Wall, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-21010; NCI-2021-10004 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-07-13; First posted 2023-08-02 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Aplastic Anemia; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Hematopoietic and Lymphoid Cell Neoplasm; Hodgkin Lymphoma; Myelodysplastic Syndrome; Myelofibrosis; Myeloproliferative Neoplasm; Non-Hodgkin Lymphoma; Plasma Cell Myeloma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anemia, Aplastic; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hematologic Neoplasms; Hodgkin Disease; Myelodysplastic Syndromes; Primary Myelofibrosis; Myeloproliferative Disorders; Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — Health Promotion; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (GO!) (Experimental): Patients undergo personalized GO! plan consisting of study visits over 50 minutes at baseline and 6 months after first visit or at the time of hospital admission for bone marrow transplant and over 25 minutes at 3 and 12 months after transplant. Patients complete questionnaires once a month for up to 6 months and wear an accelerometer for up to 6 months.
  Interventions: Other: Health Promotion and Education; Other: Medical Device Usage and Evaluation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Health Promotion and Education — Undergo GO!
Other: Medical Device Usage and Evaluation — Wear accelerometer
Other: Quality-of-Life Assessment — Complete quality of life assessments and diary entries
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This clinical trial tests whether a geriatric optimization plan (GO!) works to improve survival in patients over 60 with a hematologic malignancy or bone marrow failure syndrome eligible for allogeneic hematopoietic cell transplant. GO! focuses on creating a tailored and specific plan for each patient to make changes in their daily lives. These may include changes to their diet, sleep, activity, medicines, or even referrals to other providers depending on the patient's needs. Studying survival and quality of life in patients over 60 receiving an allogeneic hematopoietic cell transplant may help identify the effects of treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate that geriatric assessment with management (GAM) intervention will lead to improved physical functioning in allogeneic hematopoietic cell transplant (allo-HCT)-eligible older adults as measured by improvement in 6-Minute Walk Test distance of at least 35 meters.

SECONDARY OBJECTIVES:

I. To demonstrate that GAM intervention will result in improvement in Short Physical Performance Battery score by at least 1 point or score will remain >= 10 for those with baseline scores >= 10.

II. To demonstrate that GAM intervention will result in improvement in Mini Nutritional Assessment score by at least 2 points or score will remain >= 12 for those with baseline scores >= 12.

III. To evaluate change in cognition and mental health as measured by Montreal Cognitive Assessment, Personal Health Questionnaire-9, Generalized Anxiety Disorder-7, and Transplant Evaluation Rating Scale score before and after GAM intervention.

IV. To determine cumulative incidence rate for receipt of allo-HCT among study participants.

V. To measure overall survival and non-relapse mortality among study participants.

VI. To assess self-reported adherence to prescribed interventions. VII. To measure change in patient-reported quality of life immediately following GAM intervention and up to one year after completion of intervention.

EXPLORATORY OBJECTIVES:

I. To describe patterns of sleep and activity among study participants during intervention period based on accelerometer data.

II. To understand transplant physician rationale for not proceeding to allo-HCT for older patients with eligible diagnoses.

OUTLINE:

Patients undergo personalized Geriatric Optimization (GO!) plan consisting of study visits over 50 minutes at baseline and 6 months after first visit or at the time of hospital admission for bone marrow transplant and over 25 minutes at 3 and 12 months after transplant. Patients complete questionnaires once a month for up to 6 months and wear an accelerometer for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 60 years
* Diagnosed with hematologic malignancy or bone marrow failure syndrome eligible for allogeneic hematopoietic cell transplantation. This includes acute myeloid leukemia, acute lymphoblastic leukemia, myelodysplastic syndrome, myeloproliferative neoplasm, myelofibrosis, chronic myeloid leukemia, chronic lymphocytic leukemia, non-Hodgkin lymphoma, Hodgkin lymphoma, multiple myeloma, and aplastic anemia. Disease specific eligibility for allo-HCT to be determined by treating physician
* Must be able to understand written and spoken English
* Must be willing to attend all study visits and comply with study procedures for the entire length of the study

Exclusion Criteria:

* Documented history of dementia
* No possibility of proceeding to allogeneic hematopoietic cell transplant within the next 6 months as determined by treating physician
* Scheduled admission for allogeneic hematopoietic cell transplant within 30 days of enrollment
* Inability or unwillingness to give written informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in 6-Minute Walk Test distance | At 6 months before transplant, up to 12 months after transplant
  Wilcoxon signed rank test or McNemar test will be used to assess the change over time in geriatric assessment tools.

SECONDARY OUTCOMES:
Change in Short Physical Performance Battery score | At 6 months before transplant, up to 12 months after transplant
  Wilcoxon signed rank test or McNemar test will be used to assess the change over time in geriatric assessment tools.
Change in in Mini Nutritional Assessment score | At 6 months before transplant, up to 12 months after transplant
  Wilcoxon signed rank test or McNemar test will be used to assess the change over time in geriatric assessment tools.
Change in cognitive and mental health | At 6 months before transplant, up to 12 months after transplant
  Measured by Montreal Cognitive Assessment Generalized Anxiety Disorder-7. Wilcoxon signed rank test or McNemar test will be used to assess the change over time in geriatric assessment tools.
Change in cognitive and mental health | At 6 months before transplant, up to 12 months after transplant
  Measured by Personal Health Questionnaire-9. Wilcoxon signed rank test or McNemar test will be used to assess the change over time in geriatric assessment tools.
Change in cognitive and mental health | At 6 months before transplant, up to 12 months after transplant
  Measured by Generalized Anxiety Disorder-7. Wilcoxon signed rank test or McNemar test will be used to assess the change over time in geriatric assessment tools.
Change in cognitive and mental health | At 6 months before transplant, up to 12 months after transplant
  Measured by Transplant Evaluation Rating scale score. Wilcoxon signed rank test or McNemar test will be used to assess the change over time in geriatric assessment tools.
Proportion of sample achieving "normal" scores on geriatric assessment tools | At 6 months before transplant, up to 12 months after transplant
  McNemar test will be used to compare proportion of sample achieving normal scores on geriatric assessment tools.
Time to receipt of transplant | Up to 1 year after treatment
  Estimates of cumulative incidence of receipt of transplant with 95% confidence intervals will be provided for 100 days and one-year after end of treatment.
Overall survival | Up to 12 months after transplant
  Overall survival will be defined as the period from date of baseline assessment to death from any cause. Date of death will be confirmed by chart review. Will be estimated utilizing Kaplan-Meier method.
Non-relapse mortality | Up to 12 months after transplant
  Non-relapse mortality will be defined as the period from date of baseline assessment to death without evidence of relapsed primary hematologic disease. Relapse will be treated as competing risk. Documentation of date of relapse will be confirmed by chart review and collaboration with transplant physician if necessary. Estimates of cumulative incidence of non-relapse mortality with 95% confidence intervals will be provided for 100 days and one-year after end of treatment.
Adherence to prescribed geriatric optimization plan (GO!) prescription | Up to 6 months after transplant
  Will be assessed by self-report through monthly survey during intervention and at end-of-treatment assessment. Participants will be asked to estimate monthly frequency of completing all items in GO! prescription and this information will be collected through REDCap survey. Due to self-report nature of this item, no specific definition of adherence is offered beyond that which is asked of participants.
Change in quality of life | At 6 months before transplant, 3, and 6 month after transplant
  Assessed with European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire and Elderly Cancer Patients Module. Wilcoxon signed rank test or McNemar test will be used to assess the change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Wall, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu